CLINICAL TRIAL: NCT02593526
Title: Diuretic/Cool Dialysate Trial
Acronym: DIDIT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: Dialysis Clinic, Inc. (Industry)
Responsible Party: Principal Investigator, Mark Unruh, Department of Internal Medicine, Division of Nephrology Chief, University of New Mexico
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: Diuretic/Cool Dialysate Trial
Record Dates: First submitted 2015-10-20; First posted 2015-11-02 (Estimated); Results first posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2023-12

CONDITIONS: Chronic Kidney Insufficiency
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Bumetanide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- No Diuretic and 37°C dialysate (No Intervention): Standard of care, no diuretic
- No Diuretic and 35.5°C dialysate (Experimental): Cool dialysate only, no diuretic
  Interventions: Other: Cool Dialysate
- Diuretic and 37°C dialysate (Experimental): Isothermic dialysate (37°C) and bumetanide (diuretic)
  Interventions: Drug: Bumetanide
- Diuretic and 35.5°C dialysate (Experimental): Cool dialysate (35.5°C) and bumetanide (diuretic)
  Interventions: Drug: Bumetanide; Other: Cool Dialysate

INTERVENTIONS:
Drug: Bumetanide — Diuretic
  Other Names: Bumex
  Arms: Diuretic and 35.5°C dialysate; Diuretic and 37°C dialysate
Other: Cool Dialysate — Cool dialysate (35°C)
  Arms: Diuretic and 35.5°C dialysate; No Diuretic and 35.5°C dialysate

SUMMARY:
The proposed pilot study challenges the current widespread paradigm of discontinuing loop diuretics when initiating chronic HD and/or maintaining the dialysate at a constant temperature of 37 °C for all patients.

DETAILED DESCRIPTION:
This pilot/feasibility RCT will recruit for 18 months and demonstrate the feasibility and safety of performing a large scale study of diuretic use and/or cool dialysate examining recruitment, retention, and key outcomes. This study will further assess whether the use of a diuretic compared to non-use of a diuretic and/or the use of cool dialysate (35.5 ºC) compared to 37 ºC for up to 6 months will improve residual renal function (RRF), improve health reported quality of life (HRQOL) and reduce hospitalizations by randomizing 20 dialysis-naïve patients (started chronic HD in the last three months) from DCI centers in the greater Albuquerque area, to either bumetanide and cool dialysate randomized in a two-by-two factorial distribution.

ELIGIBILITY:
Inclusion Criteria:

* Primary speaking language is English.
* Patient is HD naïve (Patient may still enroll as long as no more than 12 weeks of in-center HD have been performed prior to randomization)
* HD takes place at one of the participating Dialysis Clinic Inc. (DCI) sites during the data collection period.
* Daily urine output is over 500ml.
* Patients must be willing and able to sign the consent form.

Exclusion Criteria:

* RRF <5 mL/min/1.73 m2 as determined by iohexol GFR measurement.
* Allergy or contraindication to iohexol and/or bumetanide.
* Has been undergoing dialysis for more than 12 weeks.
* Expectation that native kidneys will recover.
* History of poor adherence to treatment.
* Unable to verbally communicate in English.
* Requires more than 3 HD treatments per week due to medical co-morbidity (such as, but not limited to: severe volume overload requiring frequent HD e.g. in systemic oxalosis, or requiring total parenteral nutrition).
* Scheduled for living donor kidney transplant in the next 6 months.
* Intention to change to peritoneal dialysis, or home HD in the next 6 months.
* Plan to relocate to another center within the next 7-8 months.
* Expected geographic unavailability at a participating HD unit for >2 consecutive weeks or >4 weeks total during the next 6 months (excluding unavailability due to hospitalizations)
* Post kidney transplantation
* Currently in an acute or chronic care hospital
* Life expectancy <6 months or intention to withdraw dialysis therapy within 6 months.
* Current pregnancy
* Actively planning to become pregnant in the next 8 months
* Nursing mothers
* Current use of investigational drugs
* Participation in another non-observational clinical trial that contradicts or interferes with the therapies or measured outcomes in this trial
* Unable or unwilling to follow the study protocol for any reason (including mental incompetence)
* Unable or unwilling to provide informed consent or sign IRB-approved consent form.

The following special populations will not be included in this study:

* Patients who are too infirm or lack the capacity to meaningfully participate in medical decisions and to sign the informed consent.
* Children and adolescents constitute <2% of the dialysis population, and our preliminary survey of the study sites found no children and adolescents were active patients. In any case, the renal and other physical factors of children and adolescents with ESRD are not directly comparable to those of adults.
* Prisoners.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2022-05-27 (Actual); Study Completion 2022-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark L Unruh, MD, Principal Investigator — University of New Mexico
Locations (1):
- Dialysis Clinic Inc. - Indian School, Albuquerque, New Mexico, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from one academic medical center between December 15, 2015 and May 27, 2022, with the first participant being enrolled January 2017.
Pre-assignment Details: Of the 11 enrolled participants only 1 met randomization criteria and was randomized to treatment.
Period: Overall Study
Arm/Group | No Diuretic and 37°C Dialysate | No Diuretic and 35.5°C Dialysate | Diuretic and 37°C Dialysate | Diuretic and 35.5°C Dialysate
Started | 0 (Participants did not meet randomizations. Zero participants randomized to this arm.) | 0 (Participants did not meet randomizations. Zero participants randomized to this arm.) | 0 (Participants did not meet randomizations. Zero participants randomized to this arm.) | 1
Completed | 0 | 0 | 0 | 1
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Of the 11 enrolled participants only 1 met randomization criteria and was randomized to treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | No Diuretic and 37°C Dialysate | No Diuretic and 35.5°C Dialysate | Diuretic and 37°C Dialysate | Diuretic and 35.5°C Dialysate | Total
Number analyzed (Participants) | 0 | 0 | 0 | 1 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years |  |  |  | 0 | 0
  Between 18 and 65 years |  |  |  | 1 | 1
  >=65 years |  |  |  | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  |  |  | 0 | 0
  Male |  |  |  | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  |  |  | 0 | 0
  Asian |  |  |  | 0 | 0
  Native Hawaiian or Other Pacific Islander |  |  |  | 0 | 0
  Black or African American |  |  |  | 0 | 0
  White |  |  |  | 0 | 0
  More than one race |  |  |  | 0 | 0
  Unknown or Not Reported |  |  |  | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States |  |  |  | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Slow the Rate of Residual Renal Function (RRF)
Description: To be randomized Adequate RRF has to be determined in the first 24 hour collection (ml/min). If randomized RRF will be collected day 0 pre-dose intervention and Month 4 and 6 of intervention (3 collections) to determine if the rate was slowed. RRF is standard of care assessment for patients on dialysis for quality of life and survival.
Time Frame: 6 months
Population: Only one participant met criteria for randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | No Diuretic and 37°C Dialysate | No Diuretic and 35.5°C Dialysate | Diuretic and 37°C Dialysate | Diuretic and 35.5°C Dialysate
Number analyzed (Participants) | 0 | 0 | 0 | 1
Participants | 0 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: 7 months
Description: One participant was randomized, no adverse events were observed.
Arm/Group | No Diuretic and 37°C Dialysate | No Diuretic and 35.5°C Dialysate | Diuretic and 37°C Dialysate | Diuretic and 35.5°C Dialysate
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-07-12): https://cdn.clinicaltrials.gov/large-docs/26/NCT02593526/Prot_SAP_000.pdf
  • Informed Consent Form (2019-07-12): https://cdn.clinicaltrials.gov/large-docs/26/NCT02593526/ICF_001.pdf